CLINICAL TRIAL: NCT05978063
Title: A 2-part, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Oral Difelikefalin for Moderate-to-Severe Pruritus in Adult Subjects With Notalgia Paresthetica
Brief Title: Study to Evaluate the Efficacy and Safety of Oral Difelikefalin for Moderate to Severe Pruritus in Subjects With Notalgia Paresthetica
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: In Part A of CR845-310601, oral difelikefalin did not demonstrate a meaningful clinical benefit at any dose compared to placebo. The drug was generally well tolerated with a safety profile similar to prior trials.
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-310601
Record Dates: First submitted 2023-07-25; First posted 2023-08-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pruritus; Notalgia Paresthetica
Keywords: Notalgia Paresthetica; Pruritus; CR845; Chronic Itch; difelikefalin; Itch; Itching; Generalized pruritus; NP; Neuropathic itch
MeSH Terms: conditions — Pruritus | interventions — difelikefalin

STUDY DESIGN:
Intervention Model Description: Part A includes 4 arms and Part B includes 2 arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Difelikefalin 2.0 mg tablets (Active Comparator): Oral difelikefalin 2.0 mg tablet administered twice daily
  Interventions: Drug: difelikefalin 2.0 mg tablets
- Difelikefalin 1.0 mg tablets (Active Comparator): Oral difelikefalin 1.0 mg tablet administered twice daily
  Interventions: Drug: difelikefalin 1.0 mg tablets
- Difelikefalin 0.25 mg tablets (Active Comparator): Oral difelikefalin 0.25 mg tablet administered twice daily
  Interventions: Drug: difelikefalin 0.25 mg tablets
- Placebo tablets (Placebo Comparator): Oral placebo tablet administered twice daily
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: difelikefalin 2.0 mg tablets — Oral difelikefalin 2.0 mg administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 2.0 mg tablets
Drug: difelikefalin 1.0 mg tablets — Oral difelikefalin 1.0 mg administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 1.0 mg tablets
Drug: difelikefalin 0.25 mg tablets — Oral difelikefalin 0.25 mg administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 0.25 mg tablets
Drug: Placebo tablets — Oral Placebo administered twice daily
  Arms: Placebo tablets

SUMMARY:
This is a 2-part, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of twice-daily (BID) oral difelikefalin for moderate-to-severe pruritus in adult subjects with NP.

DETAILED DESCRIPTION:
Part A of this study will evaluate the benefit-risk of 3 doses of difelikefalin compared to placebo. The dose with the best benefit-risk profile will be further evaluated in Part B. Part A of this study comprises a 28-day Screening Period, a 7-day Run-in Period, an 8-week Double-blind Treatment Period, a 2-week Treatment Discontinuation Period, and a Safety Follow-up Visit (14 days after the last dose of study treatment).

Part B of this study will evaluate the efficacy, safety, and tolerability of oral difelikefalin. The dose of oral difelikefalin to be assessed in Part B will depend on the results of Part A. Part B of this study comprises a 28-day Screening Period, a 7-day Run-in Period, an 8-week Double-blind Treatment Period, up to a 52-week OLE Period, and a Safety Follow-up Visit.

Subjects who participated in Part A of the study may not participate in Part B.

All subjects will sign an informed consent form (ICF) and undergo screening for study eligibility.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* Subject has clinically confirmed diagnosis of active Notalgia Paresthetica;
* Subject has a history of chronic pruritus due to Notalgia Paresthetica;
* Subject has moderate to severe pruritus;
* Female subject is not pregnant or nursing during any period of the study.

Key Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Subject has pruritus attributed to a cause other than Notalgia Paresthetica;
* Subject has any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving ≥4-point improvement from baseline in the weekly mean of the daily 24-hour I-NRS score | Baseline, Week 8

SECONDARY OUTCOMES:
Proportion of subjects achieving ≥4-point improvement from baseline in the weekly mean of the daily 24-hour I-NRS score at Week 4 in Part B | Baseline, Week 4
Proportion of subjects achieving ≥4-point improvement from baseline in the weekly mean of the daily 24-hour I-NRS score at Week 2 in Part B | Baseline, Week 2
Proportion of subjects achieving ≥4-point improvement from baseline in the weekly mean of the daily 24-hour I-NRS score at Week 1 in Part B | Baseline, Week 1
Change from Baseline in the Numeric Rating Scale of Burning Sensation and Skin Tingling at Week 8 in Part B | Baseline, Week 8
Proportion of Subjects with H-IGA of Clear or Almost Clear at Week 8 in Part B | Week 8
Proportion of ≥4-point Improvement in Daily I-NRS at Day 2 in Part B | Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Cara Therapeutics, Study Director — Cara Therapeutics
Locations (57):
- United States (37):
  - Cara Therapeutics Study Site, Birmingham, Alabama
  - Cara Therapeutics Study Site, Phoenix, Arizona
  - Cara Therapeutics Study Site, Fayetteville, Arkansas
  - Cara Therapeutics Study Site, Hot Springs, Arkansas
  - Cara Therapeutics Study Site, Encino, California
  - Cara Therapeutics Study Site, Fountain Valley, California
  - Cara Therapeutics Study Site, Los Angeles, California
  - Cara Therapeutics Study Site, Northridge, California
  - Cara Therapeutics Study Site, Valencia, California
  - Cara Therapeutics Study Site, Coral Gables, Florida
  - Cara Therapeutics Study Site, Hollywood, Florida
  - Cara Therapeutics Study Site, Lutz, Florida
  - Cara Therapeutics Study Site, Margate, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Indianapolis, Indiana
  - Cara Therapeutics Study Site, Plainfield, Indiana
  - Cara Therapeutics Study Site, West Lafayette, Indiana
  - Cara Therapeutics Study Site, Baton Rouge, Louisiana
  - Cara Therapeutics Study Site, Metairie, Louisiana
  - Cara Therapeutics Study Site, New Orleans, Louisiana
  - Cara Therapeutics Study Site, Rockville, Maryland
  - Cara Therapeutics Study Site, Fort Gratiot, Michigan
  - Cara Therapeutics Study Site, Reno, Nevada
  - Cara Therapeutics Study Site, Portsmouth, New Hampshire
  - Cara Therapeutics Study Site, Verona, New Jersey
  - Cara Therapeutics Study Site, Fargo, North Dakota
  - Cara Therapeutics Study Site, Boardman, Ohio
  - Cara Therapeutics Study Site, Mason, Ohio
  - Cara Therapeutics Study Site, Pittsburgh, Pennsylvania
  - Cara Therapeutics Study Site, Charleston, South Carolina
  - Cara Therapeutics Study Site, Thompson's Station, Tennessee
  - Cara Therapeutics Study Site, Dallas, Texas
  - Cara Therapeutics Study Site, Houston, Texas
  - Cara Therapeutics Study Site, Pflugerville, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Webster, Texas
  - Cara Therapeutics Study Site, Spokane, Washington
- Canada (8):
  - Cara Therapeutics Study Site, Oakville, Ontario
  - Cara Therapeutics Study Site, Peterborough, Ontario
  - Cara Therapeutics Study Site, Richmond Hill, Ontario
  - Cara Therapeutics Study Site, Toronto, Ontario
  - Cara Therapeutics Study Site, Sherbrooke, Quebec
  - Cara Therapeutics Study Site, Montreal
  - Cara Therapeutics Study Site, Oshawa
  - Cara Therapeutics Study Site, Québec
- Germany (5):
  - Cara Therapeutics Study Site, Bad Bentheim
  - Cara Therapeutics Study Site, Berlin
  - Cara Therapeutics Study Site, Heidelberg
  - Cara Therapeutics Study Site 2, Langenau
  - Cara Therapeutics Study Site, Langenau
- Poland (5):
  - Cara Therapeutics Study Site 2, Katowice
  - Cara Therapeutics Study Site, Katowice
  - Cara Therapeutics Study Site, Sosnowiec
  - Cara Therapeutics Study Site, Szczecin
  - Cara Therapeutics Study Site, Wroclaw
- Spain (2):
  - Cara Therapeutics Study Site, Bilbao
  - Cara Therapeutics Study Site, Madrid

IPD SHARING:
Plan to Share IPD: No